CLINICAL TRIAL: NCT05747547
Title: Retinal Vascular Changes in Patients After Coronavirus Disease 2019 (COVID-19) Based on Retinal Oximetry
Brief Title: Retinal Vascular Changes in Patients After Coronavirus Disease 2019 (COVID-19)
Status: Completed | Type: Observational
Sponsor: University Hospital Olomouc (Other)
Collaborators: Palacky University (Other)
Responsible Party: Principal Investigator, Zuzana Schreiberova, Principal Investigator, University Hospital Olomouc
Other Study IDs: 9/23
Record Dates: First submitted 2023-02-24; First posted 2023-02-28 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Tonometry, Ocular; Slit Lamp Microscopy; Tomography, Optical Coherence; Angiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- mild disease: asymptomatic or paucisymptomatic patients with laboratory-confirmed severe acute respiratory syndrome coronavirus 2 infection (SARS-CoV2-infection) who received outpatient care
  Interventions: Diagnostic Test: Central visual acuity; Diagnostic Test: Intraocular pressure measurement; Diagnostic Test: Slit lamp examination; Diagnostic Test: Retinal oximetry; Diagnostic Test: Optical coherence tomography and angiography
- moderate disease: patients with laboratory-confirmed SARS-CoV2-infection and radiology-confirmed pneumonia who did not require extracorporeal membrane oxygenation
  Interventions: Diagnostic Test: Central visual acuity; Diagnostic Test: Intraocular pressure measurement; Diagnostic Test: Slit lamp examination; Diagnostic Test: Retinal oximetry; Diagnostic Test: Optical coherence tomography and angiography
- severe disease: patients with laboratory-confirmed SARS-CoV2-infection and acute respiratory distress syndrome who required extracorporeal membrane oxygenation
  Interventions: Diagnostic Test: Central visual acuity; Diagnostic Test: Intraocular pressure measurement; Diagnostic Test: Slit lamp examination; Diagnostic Test: Retinal oximetry; Diagnostic Test: Optical coherence tomography and angiography

INTERVENTIONS:
Diagnostic Test: Central visual acuity — Measurement of central visual acuity using ETDRS (Early Treatment Diabetic Retinopathy Study) optotypes or Snellen optotype chart.
Diagnostic Test: Intraocular pressure measurement — Measurement of intraocular pressure using non-contact Canon TX-20P tonometer.
Diagnostic Test: Slit lamp examination — Slit lamp examination of the anterior and posterior segment of the eye after pharmacological dilation of the pupil using application of short-time mydriatics (1% tropicamide and 10% phenylephrine).
Diagnostic Test: Retinal oximetry — Performing of retinal oximetry with an Oxymap T1 instrument (Oxymap ehf.) paired with a Topcon TRC-50DX retinal camera.
Diagnostic Test: Optical coherence tomography and angiography — Performing of optical coherence tomography and angiography with the Spectralis Optical Coherence Tomography Plus (Heidelberg Engineering).

SUMMARY:
The study examines changes in retinal oximetry in patients after COVID-19 disease. It aims to analyze and quantify possible retinal microvascular abnormalities that may result from possible post-inflammatory damage to the endothelium of the vessels associated with COVID-19 disease. Retinal vascular involvement may indicate similar changes in the vascular system in other organs.

DETAILED DESCRIPTION:
The retinal blood vessels are the only blood vessels in the body that can be observed directly. Patients with COVID-19 pneumonia have been shown to have reduced macular vessel density in the foveal region. As a result, some layers of the retina atrophy, reducing oxygen consumption by the retina. Based on this, it is expected that patients after COVID-19 pneumonia, or after a more severe course of the disease, will have normal arterial retinal oxygen saturation but higher venous retinal oxygen saturation and lower arterio-venous difference than patients after mild disease.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* history of laboratory-confirmed SARS-CoV2-infection
* transparent ocular media allowing for fundus photography
* signed informed consent

Exclusion Criteria:

* known eye disease that has been shown to affect retinal oxygen saturation (diabetic retinopathy, vascular occlusions, use of antiglaucoma drugs)
* any other serious eye disease (advanced or decompensated glaucoma, retinitis pigmentosa, age-related macular degeneration, ocular tumors)
* reduced transparency of the ocular media limiting the visualization of the ocular background and preventing a good quality image from being taken (severe dry eye syndrome, corneal scarring, cataract, significant vitreous haze, vitreous hemorrhage)
* significant refractive error not allowing for sharpening of imaging examinations
* previous intraocular surgery except cataract surgery if performed more than 3 months before the examination
* previous intravitreal application of anti-vascular endothelial growth factor therapy or laser photocoagulation of the retina
* previous severe eye injury
* acute eye infection
* known systemic disease affecting retinal oxygen saturation or causing changes in the ocular background (chronic obstructive pulmonary disease, multiple myeloma, malignant hypertension, hyperglobulinemia)
* pregnancy, breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Groups will be recruited from patients examined at the Department of Respiratory Diseases and Tuberculosis of University Hospital Olomouc at the outpatient check-up.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Successful performing of retinal oximetry images in 90% of enrolled patients. | 3 months
  90% of captured fundus images of retinal oximetry are useful for subsequent analysis.
Successful analysis of retinal oxygen saturation in 90% of enrolled patients. | 3 months
  The parameters analyzed by retinal oximetry are arterial retinal oxygen saturation (%), venous retinal oxygen saturation (%), arterio-venous difference (%), arteriolar and venular diameter (µm).

SECONDARY OUTCOMES:
Successful performing of optical coherence tomography and angiography in 90% of enrolled patients. | 3 months
  90% of captured images of optical coherence tomography and angiography are useful for subsequent analysis.
Successful analysis of optical coherence tomography in 90% of enrolled patients. | 3 months
  The parameters analyzed by optical coherence tomography are central retinal thickness (µm), ganglion cell layer thickness (µm), retinal nerve fiber layer thickness (µm), choroid thickness (µm) in the macular region and optic nerve head retinal nerve fiber layer thickness (µm).
Successful analysis of optical coherence tomography angiography in 90% of enrolled patients. | 3 months
  The parameter analyzed by optical coherence tomography angiography is the size of foveal avascular zone (µm2).

CONTACTS AND LOCATIONS:
Overall Officials: Zuzana Schreiberova, MD, Principal Investigator — University Hospital Olomouc and Palacky University Olomouc
Locations (1):
- Department of Ophthalmology, University Hospital Olomouc, Olomouc, Czechia

IPD SHARING:
Plan to Share IPD: No